CLINICAL TRIAL: NCT03608514
Title: Terlipressin Alone Versus the Standard Therapy With Catecholamines for Hepatic Patients With Septic Shock- Prospective Single Center Randomized Controlled Study.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, Eman Desoki, Fellow of intensive care medicine, NHTMRI, National Hepatology & Tropical Medicine Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NHTMRI-ICU-B
Record Dates: First submitted 2018-07-12; First posted 2018-08-01 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Resolution of Septic Shock With Terlipressin

STUDY DESIGN:
Intervention Model Description: Fifty patients will be enrolled in each arm of the study & randomly assigned in a 1:1 manner to receive either terlipressin alone versus the standard therapy (norepinephrine +/- epinephrine).
Who Masked: Participant
Masking Description: patients will be randomly assigned in 1:1 manner
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- nor-epinephrine+/- epinephrine infusion (Active Comparator): Intravenous infusion of Nor-epinephrine in an initial dose of 0.01µg/kg/min. which can be increased every 15-30 minutes to maximum 3µg/kg/min. ± intravenous infusion of epinephrine with an initial dose 0.05µg/kg/min. & can be titrated every 15-30 minutes up to 2µg/Kg/min.
  The end point is to achieve mean arterial pressure ≥ 65 mmHg & normalized lactate ≤ 2 mmol/L or lactate clearance ≥ 10% within 6 hours.
  Patients will be followed for 48 hours.
  Interventions: Drug: Experimental
- Terlipressin infusion (Other): Intravenous infusion of terlipressin by rate 1-2µg/kg/min. The end point is to achieve mean arterial pressure ≥ 65 mmHg & normalized lactate ≤ 2mmol/L or lactate clearance ≥ 10% within 6 hours.
  Patients will be followed for 48 hours.
  Interventions: Drug: Experimental

INTERVENTIONS:
Drug: Experimental — Patients in this arm of the study will receive intravenous infusion (IVi) terlipressin by rate 1-2µg/kg/min.
  Other Names: Terlipressin intravenous infusion

SUMMARY:
The purpose of this study is to evaluate the use of terlipressin compared to standard regimen in hepatic patients with septic shock. Another aim is to compare the mortality rate & the effects on renal functions in both groups.

DETAILED DESCRIPTION:
Study type:

This is a single center, prospective randomized controlled study.

Inclusion criteria:

The subjects are adults aged between 18 & 70 years who will be admitted to the intensive care unit (ICU) of National Hepatology & Tropical Medicine Research Institute (NHTMRI).

All patients that will be included in the study should have septic shock diagnosed by having sepsis with an underlying circulatory and cellular/metabolic abnormality

Exclusion criteria:

Patients will be excluded if they are pregnant, have uncontrolled hypertension, ischemic skin necrosis, present or suspected coronary artery disease, present or suspected acute mesenteric ischemia, or peripheral vascular diseases (e.g. Raynaud's syndrome or related diseases) or hypersensitivity to terlipressin.

Study design:

Fifty patients will be enrolled in each arm of the study & randomly assigned in a 1:1 manner to receive either intravenous infusion (IVi) terlipressin by rate 1-2µg/kg/min. or intravenous infusion norepinephrine in an initial dose of 0.01µg/kg/min which can be increased every 15-30min. to 3µg/kg/min. maximum ± epinephrine with an initial dose 0.05µg/kg/min. IVi & can be titrated every 15-30min. The increments of epinephrine dose will be 0.05- 0.2µg/kg/min. and up to 2µg/Kg/min. The end point of the study will be achieving mean arterial pressure ≥ 65mmHg & normalized lactate ≤ 2mmol/L or lactate clearance ≥ 10% within 6hours All demographic data will be obtained at time of admission, including the patients' age, sex, body mass index (BMI), associated co-morbidities (diabetes mellitus, hypertension), Child-Pugh score and Sequential Organ Failure Assessment (SOFA).

Vital signs including the heart rate, mean arterial pressure (MAP) through arterial cannula, central venous pressure (CVP) through a catheter inserted either in the internal jugular vein or the subclavian vein will be measured at admission and at regular intervals. The volume & fluid balance will be recorded at admission and then will be followed up daily and recorded as required. Daily ECG with ST analysis, lactate level & ScVO2 will be measured on admission and then recorded at regular intervals during treatment after 2, 6, 12, 24 & 48hours.

Organ dysfunction and injury (aspartate aminotransferase, alanine amino-transaminase, total bilirubin, international normalized ratio, serum creatinine and troponin-I) will be analyzed at admission, and after 12, 24 & 48hours of treatment.

The rate of norepinephrine ± epinephrine infusion as well as terlipressin dose required to keep MAP at 65 mmHg will be recorded at baseline and 6, 12, 24, and 48hours after treatment.

Twenty-eight day mortality will be followed by phone calls to the patient or one of his/her first-degree relatives.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 & 70years who will be admitted to the intensive care unit (ICU) of National Hepatology & Tropical Medicine Research Institute (NHTMRI).

All patients that will be included in the study should have septic shock diagnosed by having sepsis with an underlying circulatory and cellular/metabolic abnormality.

Exclusion Criteria:

* Patients will be excluded if they are pregnant, have uncontrolled hypertension, ischemic skin necrosis, present or suspected coronary artery disease, present or suspected acute mesenteric ischemia, or peripheral vascular diseases (e.g. Raynaud's syndrome or related diseases) and hypersensitivity to Terlipressin.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic stability & optimization; mean blood pressure more than or equal 65mmHg | 48hours up to 7days
  how fast hemodynamic stability will be achieved in each arm of the study
mortality | 28 days
  28-day mortality will be followed by phone calls to the patient or one of his/her first degree relatives
Hemodynamic stability & optimization; mean blood pressure | 48hours up to 7days
  for how long hemodynamic stability will be maintained
Hemodynamic stability & optimization, lactate clearance to be 2mmol/L | 48hours up to 7days
  how fast it will be achieved

CONTACTS AND LOCATIONS:
Locations (1):
- NHTMRI, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol